CLINICAL TRIAL: NCT00072033
Title: Docetaxel and Cisplatin Chemo- and Radiochemotherapy Followed by Surgery in Patients With Locally Advanced Esophageal Cancer - A Multicenter Phase II Trial
Brief Title: Neoadjuvant Docetaxel and Cisplatin Plus Chemoradiotherapy Followed By Surgery in Treating Patients With Locally Advanced, Resectable Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 75/02; EU-20323
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Esophageal Cancer
Keywords: stage II esophageal cancer; stage III esophageal cancer; adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Active Comparator): Docetaxel and Cisplatin chemo- and radiochemotherapy followed by surgery
  Interventions: Drug: Cisplatin and Docetaxel

INTERVENTIONS:
Drug: Cisplatin and Docetaxel — cisplatin and docetaxel chemo- and radiochemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and cisplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving combination chemotherapy with radiation therapy before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well giving docetaxel and cisplatin together with chemoradiotherapy followed by surgery works in treating patients with locally advanced, resectable esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effectiveness of neoadjuvant docetaxel and cisplatin and chemoradiotherapy followed by surgery, in terms of pathological response rate, in patients with locally advanced, resectable esophageal cancer.
* Determine the feasibility of this regimen, in terms of successful completion of therapy and survival at 30 days postoperatively, in these patients.

Secondary

* Determine the parameters of disease control in these patients and toxicity of this regimen and compare these parameters with published results.
* Correlate early improvement of dysphasia after 1-2 courses of chemotherapy with predictive value with regard to tumor response and long-term disease control in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the clinical benefit of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Neoadjuvant chemotherapy: Patients receive docetaxel IV over 1 hour and cisplatin IV over 1 hour on days 1 and 22.
* Chemoradiotherapy: Beginning 21 days after the last dose of neoadjuvant chemotherapy, patients receive docetaxel IV over 30 minutes and cisplatin IV over 1 hour once a week and undergo radiotherapy 5 days a week for 5 weeks.
* Surgery: Patients undergo surgery 3-8 weeks after the final administration of radiotherapy.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, day 22 of chemotherapy, day 1 of chemoradiotherapy, before surgery, and then every 3 months for 1 year.

Patients are followed every 3 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 22-66 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the thoracic esophagus, including the gastroesophageal junction (Siewert type I)

  * Locally advanced disease that is technically operable with curative intent (R0)
  * T3, N0 OR T1-3, N+ OR T4, NX
  * No T1-2, N0
  * No inoperable T4 (unequivocal organ involvement)
  * No distant metastasis, including M1a lymph node status

    * Lymph nodes suspicious of M1a status by CT scan, PET scan, or ultrasound must be verified by fine-needle aspiration cytology
* No carcinoma of the cervical esophagus
* Obstructive tumors allowed

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* AST no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* Bilirubin no greater than 1.5 times ULN

Renal

* Creatinine clearance greater than 60 mL/min

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No unstable angina pectoris
* No myocardial infarction within the past 3 months
* No significant arrhythmias
* No other severe or uncontrolled cardiovascular disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after study treatment
* No definite contraindications to corticosteroids as premedication
* No geographic situation that would preclude proper staging and follow-up
* No active uncontrolled infection
* No preexisting peripheral neuropathy greater than grade 1
* No uncontrolled diabetes mellitus
* No active autoimmune disease
* No other serious medical condition that would preclude study participation
* No other prior or concurrent malignancy except nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix
* No significant neurologic or psychiatric disorder, including psychotic disorders, dementia, or seizures that would preclude comprehension and ability to provide informed consent and complete quality of life questionnaires

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the chest

Surgery

* Not specified

Other

* More than 30 days since prior treatment on another clinical trial
* No other concurrent experimental drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-03; Primary Completion 2003-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of successful study therapy completion and survival after surgery | 30 days

SECONDARY OUTCOMES:
Adverse events | 30 days
Overall survival | Life-long
Feasibility in Switzerland after surgery | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ruhstaller, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (9):
- Switzerland (9):
  - Kantonspital Aarau, Aarau
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Spitaeler Chur AG, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale Civico, Lugano
  - Kantonsspital - St. Gallen, Sankt Gallen
  - City Hospital Triemli, Zurich

REFERENCES:
- [Result] Jost C, Binek J, Schuller JC, Bauerfeind P, Metzger U, Werth B, Knuchel J, Frossard JL, Bertschinger P, Brauchli P, Meyenberger C, Ruhstaller T. Endosonographic radial tumor thickness after neoadjuvant chemoradiation therapy to predict response and survival in patients with locally advanced esophageal cancer: a prospective multicenter phase ll study by the Swiss Group for Clinical Cancer Research (SAKK 75/02). Gastrointest Endosc. 2010 Jun;71(7):1114-21. doi: 10.1016/j.gie.2009.12.015. Epub 2010 Mar 20. PMID 20304399
- [Result] Klaeser B, Nitzsche E, Schuller JC, Koberle D, Widmer L, Balmer-Majno S, Hany T, Cescato-Wenger C, Brauchli P, Zund M, Pestalozzi BC, Caspar C, Albrecht S, von Moos R, Ruhstaller T. Limited predictive value of FDG-PET for response assessment in the preoperative treatment of esophageal cancer: results of a prospective multi-center trial (SAKK 75/02). Onkologie. 2009 Dec;32(12):724-30. doi: 10.1159/000251842. Epub 2009 Nov 9. PMID 20016233
- [Result] Ruhstaller T, Widmer L, Schuller JC, Roth A, Hess V, Mingrone W, von Moos R, Borner M, Pestalozzi BC, BalmerMajno S, Koberle D, Terraciano L, Schnider A, Bodis S, Popescu R; Swiss Group for Clinical Cancer Research (SAKK). Multicenter phase II trial of preoperative induction chemotherapy followed by chemoradiation with docetaxel and cisplatin for locally advanced esophageal carcinoma (SAKK 75/02). Ann Oncol. 2009 Sep;20(9):1522-1528. doi: 10.1093/annonc/mdp045. Epub 2009 May 22. PMID 19465425
- [Result] Schuller JC, Balmer-Majno S, Mingrone W, et al.: Preoperative induction chemotherapy with docetaxel-cisplatin followed by concurrent docetaxel-cisplatin and radiation therapy (RT) in patients with locally advanced esophageal cancer: final results of the multicenter phase ll trial SAKK 75/02. [Abstract] J Clin Oncol 26 (Suppl 15): A-4550, 2008.
- [Result] Ribi K, Nitzsche E, Schuller J, et al.: PET scanning and patient reported dysphagia before and after chemotherapy (CT) for prediction of pathological response after CT and chemoradiotherapy (CRT) in patients with locally advanced esophageal cancer (EC): a multicenter phase ll trial of the Swiss. [Abstract] J Clin Oncol 25 (Suppl 18): A-4587, 2007.
- [Result] Ruhstaller T, Widmer L, Majno SB, et al.: Preoperative induction chemotherapy with docetaxel-cisplatin followed by concurrent docetaxel-cisplatin and radiation therapy in patients with locally advanced esophageal cancer: a prospective, multicenter phase ll trial of the Swiss Group for Clinical Cancer Research. [Abstract] J Clin Oncol 25 (Suppl 18): A-4562, 2007.
- [Derived] Steffen T, Dietrich D, Schnider A, Kettelhack C, Huber O, Marti WR, Furrer M, Gloor B, Schiesser M, Thierstein S, Brauchli P, Ruhstaller T; Swiss Group for Clinical Cancer Research (SAKK). Recurrence Patterns and Long-term Results After Induction Chemotherapy, Chemoradiotherapy, and Curative Surgery in Patients With Locally Advanced Esophageal Cancer. Ann Surg. 2019 Jan;269(1):83-87. doi: 10.1097/SLA.0000000000002435. PMID 28742685